CLINICAL TRIAL: NCT03975101
Title: Autologous Very Small Embryonic-like Stem Cells(VSELs) for Knee Osteoarthritis
Brief Title: Very Small Embryonic-like Stem Cells for Knee Osteoarthritis
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Policy changes have contributed to the failure to carry out smoothly
Sponsor: Fuda Cancer Hospital, Guangzhou (Other)
Collaborators: Guangzhou Four-Leaf Clover HealthTech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VSEL-knee
Record Dates: First submitted 2019-05-31; First posted 2019-06-05 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-05

CONDITIONS: Stem Cell Transplant Complications; Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Three experimental groups were injected with different doses of VSEL, and the control group was injected with platelet-containing serum that dissolved VSEL.
Who Masked: Investigator
Masking Description: The investigators screen patients with similar knee condition to ensure a small difference, and they randomized different numbers of VSELs to the patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- VSEL Max (Experimental): A mean volume of 5.5 mL platelet-rich plasma containing approximately 120,000 cells were prepared and injected into the selected knee of the patient
  Interventions: Biological: very small embryonic-like stem cell
- VSEL Medium (Experimental): A mean volume of 5.5 mL platelet-rich plasma containing approximately 90,000 cells were prepared and injected into the selected knee of the patient
  Interventions: Biological: very small embryonic-like stem cell
- VSEL Mini (Experimental): A mean volume of 5.5 mL platelet-rich plasma containing approximately 60,000 cells were prepared and injected into the selected knee of the patient
  Interventions: Biological: very small embryonic-like stem cell
- Control (No Intervention): A mean volume of 5.5 mL platelet-rich plasma containing no VSELs injected into the selected knee of the patient

INTERVENTIONS:
Biological: very small embryonic-like stem cell — Mononuclear cells were collected from peripheral blood of each patient using a machine, VSELs were isolated, and each group was injected according to different numbers after activation
  Other Names: VSEL
  Arms: VSEL Max; VSEL Medium; VSEL Mini

SUMMARY:
The aim of this study is the safety and efficacy of autologous very small embryonic-like stem cells(VSELs) to knee osteoarthritis.

DETAILED DESCRIPTION:
VSELs come from the patient's peripheral blood, and will be injected in the most painful knee, or the worse knee on physical examination. Then follow-up the knee pain and imaging changes at 6 months and 1 year after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients had moderate to severe osteoarthritis of both knees.
* Those had mechanical pain of knee joints, which was aggravated by walking or stair climbing.
* Those complained of gelling pain of knee joint.
* Those have crepitus and limitation of the joint range of motion with joint bony hypertrophy on physical examination, X-rays showed narrowing of joint space and osteophyte formation

Exclusion Criteria:

* Diabetic foot and patients with obvious edema in the legs caused by various causes
* Blood disease patients, thrombocytopenia or dysfunction, hypofibrinemia or anticoagulant therapy, long-term use of aspirin

Ages: 50 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2019-07-05 (Actual); Primary Completion 2020-05-25 (Estimated); Study Completion 2020-06-15 (Estimated)

PRIMARY OUTCOMES:
Change of knee pain score | 2-4 weeks after injection
  Pain assessment by visual analogue score (VAS). 0 point: no pain; 1-3 points: there is a slight pain that can be tolerated; 4-6 points: the patient has pain and affects sleep, and can still bear it; 7-10 points: the patient has progressively strong pain, pain is unbearable, affecting appetite and sleep

SECONDARY OUTCOMES:
Change of knee pain score | 6 months after injection
  Pain assessment by visual analogue score (VAS). 0 point: no pain; 1-3 points: there is a slight pain that can be tolerated; 4-6 points: the patient has pain and affects sleep, and can still bear it; 7-10 points: the patient has progressively strong pain, pain is unbearable, affecting appetite and sleep
Imaging changes in the knee joint | 6 months after injection
  Magnetic resonance image (MRI) examination of the smoothness of the knee joint surface, ligament, soft tissue and meniscus damage
Change of knee pain score | 12 months after injection
  Pain assessment by visual analogue score (VAS). 0 point: no pain; 1-3 points: there is a slight pain that can be tolerated; 4-6 points: the patient has pain and affects sleep, and can still bear it; 7-10 points: the patient has progressively strong pain, pain is unbearable, affecting appetite and sleep
Imaging changes in the knee joint | 12 months after injection
  MRI examination of the smoothness of the knee joint surface, ligament, soft tissue and meniscus damage

CONTACTS AND LOCATIONS:
Locations (1):
- Biological treatment center in Fuda cancer hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No